CLINICAL TRIAL: NCT02578615
Title: Physiotherapie Bei Chronischer Metatarsalgie - Ein Vergleich Klinischer Parameter Vor Und Nach Therapie gemäß Spiraldynamik®- Konzept
Brief Title: Physiotherapy for Chronic Metatarsalgia
Status: Completed | Type: Observational
Sponsor: Spiraldynamik AG (Other)
Responsible Party: Principal Investigator, Dr.Albers, Gertraud, Dr. med., Spiraldynamik AG
Other Study IDs: 2014-0528
Record Dates: First submitted 2015-10-13; First posted 2015-10-19 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Metatarsalgia
MeSH Terms: conditions — Metatarsalgia | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: physiotherapy — physiotherapeutic intervention according to the principles of the Spiraldynamik® concept

SUMMARY:
The pilot study was conducted in the form of an open prospective single-arm observational study with 28 patients who received physiotherapy at the Spiraldynamik® Med Center in Zurich.

DETAILED DESCRIPTION:
The pilot study was conducted in the form of an open prospective single-arm observational study. The data of 28 patients who received physiotherapy at the Spiraldynamik® Med Center in Zurich was evaluated. The endpoints of Visual Analog Scale Foot and Ankle (VAS FA), Activity Index (AI), plantar and inter-metatarsal pres-sure pain, rearfoot angle and dorsal extension capability of the upper ankle joint were individually compared and analyzed before and after therapy.

ELIGIBILITY:
Inclusion Criteria:

* main diagnosis: Metatarsalgia
* secondary diagnosis: Hallux rigidus,Hallux valgus, Knick-Senk-Spreizfuß, Hohlfuß
* age 30-75 Jahre, gender both
* chronic ( ≥ 3 month),
* pain ≥ 1 visuell analog scale (VAS)
* no other complementary therapy

Exclusion Criteria:

* local: trauma, fracture, tumore, infectionen
* pain after forefoot - operation
* neurological diseases
* generell: somatoform, pension covet

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic metatarsalgia
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2013-12; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale Foot and Ankle (VAS FA) | 9 weeks

SECONDARY OUTCOMES:
Activity Index (AI) | 3, 8 weeks
plantar and inter-metatarsal pressure pain - measured dichotom | 9 weeks
  measured dichotom - pain triggered or not
rearfoot angle measured in degree ° | 9 weeks
  measured in degree, during standing: the angle for pes valgus (measured at the position of calcaneus)
dorsal extension capability of the upper ankle joint measured in degree ° | 9 weeks